CLINICAL TRIAL: NCT00379119
Title: Androgen Blockade Therapy and Thymic Function in Individuals Over 50 Years of Age With Adenocarcinoma of the Prostate: A Cross-Sectional Study
Brief Title: Effect of Androgen Blockade Therapy on Thymus Function in Older Patients Who Have Undergone Radical Prostatectomy for Localized Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000455646; UCSF-035511
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis
Other: flow cytometry
Other: physiologic testing
Procedure: computed tomography

SUMMARY:
RATIONALE: Studying changes in thymus function in patients who have been undergoing androgen blockade therapy for prostate cancer may help doctors learn more about how well patients will respond to treatment, may help in planning cancer treatment, and may help the study of cancer in the future.

PURPOSE: This clinical trial is studying the effect of androgen blockade therapy on thymus function in older patients who have undergone radical prostatectomy for localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if inhibition of sex steroid action is associated with increased thymic size in older patients who have undergone radical prostatectomy for localized adenocarcinoma of the prostate.
* Determine if inhibition of sex steroid action is associated with an increase in the absolute number or percentage of circulating "naive" phenotype T cells, and/or an increase in the frequency of T-cell receptor excision circles in peripheral blood cells.

OUTLINE: This is a nonrandomized, single-blind, cohort study. Patients are stratified according to hormonal therapy after surgery (yes vs no).

Patients undergo CT scan of the thymus. Blood samples are analyzed by flow cytometry to determine phenotype of T cells.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Underwent prior radical prostatectomy as local definitive therapy for prostate cancer
* Meets criteria for 1 of the following strata:

  * Has received ≥ 9 months of androgen blockade therapy (either single-agent luteinizing hormone-releasing hormone or combined androgen blockade) for serologic progression after surgery

    * Serologic progression defined as a rising prostate-specific antigen, which has risen serially on two determinations (from baseline) ≥ 1 week apart, and no objective evidence of metastatic disease
    * Prior radiotherapy for serologic progression allowed
  * Did not receive any form of androgen blockade therapy within the past 9 months
* No metastatic disease by abdominal/pelvic CT scan and whole-body scan

PATIENT CHARACTERISTICS:

* Able to tolerate CT scanning in the supine position
* No prior medical condition known to have effects on the thymus, including myasthenia gravis, lymphoma, hyperthyroidism, or cachexia
* No autoimmune disorders
* No acute illness, including active infection requiring antibiotics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy
* No prior immunological therapy
* No prior single-agent antiandrogen (e.g., high-dose bicalutamide)
* No prior or concurrent 5-alpha reductase inhibitors (e.g., finasteride), PC-SPES, or estrogen-containing nutraceuticals
* No concurrent systemic steroid therapy (topical steroids allowed)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals >50 years of age with prostate cancer
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Size of thymus as assessed by CT scan | approximately 4 hours during one session
Fraction and absolute number of circulating peripheral blood CD4+ and CD8+ T cells with a "naive" phenotype | approximately 4 hours during one session
Number of T-cell receptor excision circles in peripheral blood cells | approximately 4 hours during one session

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. McCune, MD, PhD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States